CLINICAL TRIAL: NCT06446921
Title: The Effect of a Ginger Formulation Supplementation on Gastrointestinal Complaints in Healthy Adults: A Randomized, Doubleblind, Placebo Controlled Trial
Brief Title: The Effect of a Ginger Supplement on Digestive Complaints in Healthy Adults Versus a Placebo
Acronym: GIGI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Givaudan France Naturals (Industry)
Collaborators: Analyze & Realize (Network); University Hospital of Leuven Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GIV/010123
Record Dates: First submitted 2024-05-23; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Dyspepsia
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Intervention Model Description: randomized placebo controlled double blind trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ginger formula (Experimental): 100 mg of ginger formula per capsule 2 capsules per day during 8 weeks
  Interventions: Dietary Supplement: Ginger formula
- Placebo formula (Placebo Comparator): 2 capsules per day during 8 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ginger formula — supplement delivering a minimum of 20 mg of gingeroids / d
  Arms: Ginger formula
Dietary Supplement: Placebo — arabic gum
  Arms: Placebo formula

SUMMARY:
The aim of this clinical study is to investigate the effect of a ginger formulation as a dietary supplement on gastrointestinal complaints in healthy adults.

The effect of this formula will be compared to a placebo after 8 weeks of consumption.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-65 years
* Body Mass Index (BMI) 18.5 - 30.0 kg/m2 (limits included)
* Otherwise healthy subjects with Postprandial Distress Syndrome (PDS) as defined by ROME IV criteria: Must include one or both of the following criteria* at least 3 days a week: - Bothersome postprandial fullness (i.e. severe enough to impact on usual activities)
* Bothersome early satiation (i.e. severe enough to prevent finishing a regular size meal)

  *Criteria fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis with no apparent evidence of organic, systemic or metabolic disease or structural disease by standard clinical examination by the investigator at V0 that is likely to explain the complaints
* Documented Helicobacter pylori negative subjects according to a validated previous test (histological, breath, stool antigen or serological test) in the last 5 years or if not, with a rapid assay realized during V0
* Negative urine pregnancy test for women in childbearing age at V0 At V1, after 1-week diary completion, mean "PDS score" on LPDS scale ≥ 1 and <3 (mild and moderate) As per this randomization criterion, any subjects with a "PDS score" of ≥3 (severe or very severe) or <1 (too low) at V1 will be withdrawn from the study.

For assessment of PDS, the last 7 consecutive days before V1 should be used to calculate the score.

Exclusion Criteria:

* Subjects with dominant Epigastric Pain Syndrome (EPS) (as per Rome IV criteria) as main complaints at V0 as per investigator's judgement
* Subject with a dominant Irritable Bowel Syndrome (IBS) as per Rome IV criteria at V0 as per investigator's judgement
* Subjects suffering from or with history of dominant gastroesophageal reflux disease (GERD)-like symptoms at V0 as per investigator's judgement
* Self-reported organic findings in endoscopy in the last 5 years (if any) likely to explain dyspeptic symptoms
* Subject with other chronic gastrointestinal (GI) disorders (e.g. inflammatory bowel disease, coeliac disease)
* History of major gastrointestinal surgery (except for appendectomy or cholecystectomy)
* Suffering from or history of severe chronic disease in the last 5 years (e.g. cancer, HIV, hepatic or biliary disorders ongoing, pancreatic disease, kidney disease, uncontrolled cardiovascular disease, or chronic respiratory diseases) (self-reported)
* Presence of an organic cause explaining the dyspeptic complaints (e.g. peptic ulcer disease or parasitic infection) (self-reported)
* Family history of oesophageal or gastric cancer
* Subjects with diabetes (self-reported)
* Subjects with PHQ-9 (PATIENT HEALTH QUESTIONNAIRE)(score over 15 at V0
* Subjects with GAD-7 (Generalized Anxiety Disorder 7-item) score over 15 at V0
* Active psychiatric conditions (stable dose of 1 antidepressant is allowed, no other medication for psychiatric conditions)
* Subjects under treatment for dyspepsia complaints such as Proton Pump Inhibitors (PPI), Histamine 2 receptor antagonists (H2RAs), prokinetics, within the last 6 weeks before V0 and during the study and not willing to refrain their use during the study
* Subjects under opioids or immunosuppressants (antihistaminics and topical corticosteroids (nasal sprays, cutaneous) are allowed) or Non-steroidal anti-inflammatory drugs (NSAIDS) within the last 2 weeks before V0 and during the study and not willing to refrain their use during the study
* Subjects under treatment of antibiotics within the last 2 months before V0
* Subjects accustomed to use an anti-acid more than 3 times a week and not willing to refrain any consumption of these during the study
* Subjects under treatment of systemic corticoids within the last 3 months before V0 and not willing to refrain their use during the study
* Recent gastroenteritis or food borne illness such as confirmed food poisoning within the last 1 month before V0
* Under dietary supplement or treatment which could significantly affect parameters followed during the study according to the investigator (i.e. with laxative effect, with antidiarrheal effect, containing plant extracts (including ginger extracts), any formulation for digestive health, probiotics, prebiotics, symbiotic, vitamins and minerals) within the last 6 weeks before V0 or not willing to refrain from their consumption during the study
* Subjects used to consume any food and/or drink and/or condiment containing ginger (gari, pickled ginger, Japanese food, tea or infusion…) defined as more than 4 times a week before the study
* Subjects who do not agree to limit any ginger consumption during the study to maximally 4 times a week during the study
* With a known or suspected food allergy or intolerance or hypersensitivity to any of the study products' ingredients and/or for the subgroup (with the gastric emptying test) to any components of the standard meals
* Pregnant or breastfeeding females, or wishing to become pregnant during the study
* With significant change of dietary habits or trying to lose weight within the last 3 months before V0 or planning to change dietary habits during the study or with eating disorders as per investigator judgement
* Following any specific diet such as high-protein, vegan, hypocaloric, ketogenic diet low in FODMAPs (Fructo-, Oligo, Di-Monosaccharides, And Polyols) except for vegetarian which is allowed
* Any change in the physical activity within the last 3 months before V0 or planning to change during the study or participant near or in the peak of training for an athletic race or competition
* Ongoing abuse of drugs, alcohol and / or medication at V0 or history of substance abuse within the last 12 months before V0
* Drinking more than 2 glasses of alcohol per day, every day and without interruption
* Smoking > 10 cigarettes per day
* Heavy caffeinated beverage consumption (>400 mg caffeine/day, i.e. more than 3 mugs of filter coffee or 4 espressos) within the last 2 weeks before V0 and during the study
* Any reason or condition that in the judgment of the clinical investigator(s) may put the subject at unacceptable risk or that may preclude the subject from understanding or complying with the study's requirements
* Participation in any other clinical trial within the last 30 days before V0 and during the study
* Clinically relevant deviations from safety laboratory parameters (see section 11.8.3)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Leuven Postprandial Distress scale (LPDS) | daily, up to 66 days after the day of inclusion. from the day after inclusion until 8 weeks after randomization visit
  The LPDS is a questionnaire consisting of eight items: early satiation, postprandial fullness, upper abdominal bloating, epigastric pain, epigastric burning, nausea, belching and heartburn. Each symptom will be rated on a 5-point Likert-type scale: absent=0, mild=1, moderate=2, severe=3 and very severe=4 over a period of one day.

SECONDARY OUTCOMES:
Short Form Nepean Dyspepsia Index (SF-NDI) | monthly, from the day of randomization visit (V1) till end of study visit (V3) after 2 months
  The Short Form (SF) Nepean Dyspepsia Index is a 10-item questionnaire with 5 sub-scales each examining the influence of dyspepsia on domains of health in subjects, namely tension/anxiety, interference with daily activities, disruption to regular eating/drinking, knowledge towards/control over disease symptoms and interference with work/study, with each sub-scale containing two items. Each item is measured by a 5-point Likert scale ranging from 0 (not at all or not applicable), 1 (a little), 2 (moderately), 3 (quite a lot) to 4 (extremely) scores.
Overall Treatment Effect (OTE) | monthly, from the day of randomization visit (V1) till end of study visit (V3) after 2 months
  Subjects instructed to answer the question: "How were your gastric symptoms during the past week in comparison with the baseline period preceding the intake of the food supplement? " (7 point Likert scale)
Gastric emptying | twice : basal at visit V1 (randomization) and after 2 months
  The gastric emptying breath test is a standard tool to measure gastric emptying rate in subjects with dyspeptic symptoms. After eating, subjects will provide a breath sample and will score the severity (0: absent - 4: very severe) of 6 epigastric symptoms (fullness, bloating, nausea, epigastric pain, burning, and belching) every 15 minutes until 4 hours postprandially.
Chalder fatigue scale | monthly, from the day of randomization visit (V1) till end of study visit (V3) after 8 weeks
  Each of the 11 items are answered on a 4-point scale ranging from asymptomatic to maximum symptomatology. Using the Likert scoring method, responses on the extreme left receive a score of 0, increasing to 1, 2 or 3 as they become more symptomatic. The respondent's global score can range from 0 to 33. The global score also spans two dimensions-physical fatigue (measured by items 1-7) and psychological fatigue (measured by items 8-11). The Likert scoring system allows for means and distributions to be calculated for both the global total as well as the two sub-scales.
Perceived stress scale (PSS-10) | monthly, from the day of randomization visit (V1) till end of study visit (V3) after 2 months
  The PSS-10 is a self-questionnaire comprising 10 items and allowing each item to be evaluated on its frequency of occurrence during the previous month using a 5-point scale ranging from 0 = never to 4 = very often (Cohen & Williamson, 1988; Bellinghausen, 2009). The PSS-10 consists of 10 items from the PSS-14 (items 1, 2, 3, 6, 7, 8, 9, 10, 11, and 14). The PSS-10 allows the assessment of perceived stress without any loss of psychometric quality.
  PSS-10 scores are obtained by reversing responses (e.g., Never = 4, Almost Never = 3, Sometimes = 2, Fairly Often = 1, Very Often= 0) to the four positively stated items (items 4, 5, 7 and 8 from the PSS-10, corresponding to items 6, 7, 9 and 10 from the original PSS-14) and then summing across all scale items.
  Individual scores on the PSS-10 can range from 0 to 40 with higher scores indicating higher perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Vanuytsel, Pr, Principal Investigator — UZ Leuven